CLINICAL TRIAL: NCT06526533
Title: Generating New Evidence to Reduce Major Complications to Improve the Safety and Efficacy of ECMO in Severe Cardiac and Respiratory Failure (RECOMMEND)
Brief Title: RECOMMEND Platform Trial
Acronym: RECOMMEND
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Monash University (Other); Berry Consultants (Other); Research Path (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ANZIC-RC/CH006
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; ARDS (Acute Respiratory Distress Syndrome); Intensive Care Medicine; Cardiac Arrest (CA); Critical Illness
Keywords: ECMO; ICU; Platform Trial; Australia; Cardiac; Respiratory; VA; VV; eCPR; Adaptive
MeSH Terms: conditions — Acute Lung Injury; Heart Arrest; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group/Arm (Other): RBC Transfusion Domain:
  Patients on ECMO in ICU enrolled in the RBC Transfusion Domain of RECOMMEND. Patients receive one of two RBC transfusion strategies (restrictive or liberal)
  Interventions: Other: Liberal RBC Transfusion; Other: Restrictive RBC Transfusion

INTERVENTIONS:
Other: Liberal RBC Transfusion — Liberal transfusion trigger group (patient receives RBC transfusion if Hb <90g/L).
Other: Restrictive RBC Transfusion — Restrictive transfusion trigger group (patient receives RBC transfusion if Hb <70g/L).

SUMMARY:
The goal of this platform trial is to determine the efficacy, safety and cost-effectiveness of various interventions in patients with acute cardiorespiratory failure requiring extracorporeal membrane oxygenation (ECMO)

The main question the platform trial aims to address is to determine the effect of a range of interventions on survival, organ support and resource utilisation to day 28 for hospitalised patients receiving ECMO.

Researchers will compare various interventions within multiple platform trial domains to see if the interventions have effects on survival, organ support and resource utilisation for the patient cohort.

Participants will be enrolled in accordance with the platform trial's domain structure to answer the research questions.

DETAILED DESCRIPTION:
The RECOMMEND Platform trial is an investigator initiated, multicentre, open labelled, randomised controlled Platform Trial that will utilise Bayesian adaptive logic to investigate the efficacy and safety of multiple study interventions simultaneously or sequentially in cohorts of adult patients who are receiving ECMO from ICUs participating in the national ECMO registry (EXCEL) in Australian hospitals (EXCEL Registry NCT03793257).

In this platform trial, various interventions will be investigated for their potential to improve outcomes for patients undergoing ECMO.

Extracorporeal Membrane Oxygenation (ECMO) is an invasive and resource intensive treatment used to support critically ill patients suffering from severe cardiac arrest, cardiac failure or respiratory failure. ECMO provides mechanical circulatory support, temporarily replacing the function of the heart and/or lungs, allowing time for these organs to recover.

Globally, the use of ECMO has increased rapidly over the past decade. It is both invasive and expensive, with the average cost for a single admission in Australia exceeding more than $180,000 and a total annual cost of > $75 million. Despite its high cost, ECMO is associated with a high mortality rate, and many survivors have compromised functional recovery for months or years after discharge from hospital, further adding to the long-terms costs of care.

The main complications reported in the national ECMO registry from 2019-2022 include bleeding (51.4%), renal failure and fluid overload (78.4%), and death and ongoing disability (66%). These were confirmed as research priorities by consumers and end-users. While the use of ECMO increases swiftly, the evidence base to support the growing patient numbers receiving this care has not grown at the same rate, resulting in important evidence gaps.

The RECOMMEND Platform Trial will address these evidence gaps in ECMO services in Australia. A platform trial is a type of study design that evaluates multiple treatment interventions for a single condition or device simultaneously within a single, overarching framework. This framework operates similarly to a standard operating procedure for study logistics, ethics management, funding, staffing, and statistical and data collection methods. Having an approved process (platform) for the 'Platform Trial' to operate saves time and money and increases speed of clinical trial onboarding to outcome resolution for researchers, hospital staff, ethics committees, and stakeholders. With this platform in place, future studies of similar ECMO outcomes can be onboarded more efficiently, as described above, and it creates a more powerful pool of data for impactful patient-centred research.

Over the lifetime of RECOMMEND, it is anticipated that new interventions will be added as new domains. The creation of new domains will be considered according to priorities set by relevant working groups, based on existing or new clinical need and there being sufficient statistical power available within RECOMMEND.

ELIGIBILITY:
PLATFORM INCLUSION CRITERIA:

* Patients receiving ECMO
* Patients enrolled in the EXCEL Registry - NCT03793257

PLATFORM EXCLUSION CRITERIA:

* Treating clinician regards death as imminent and inevitable
* Treating clinician determines it is not in the patient's best interests

RBC TRANSFUSION DOMAIN INCLUSION CRITERIA:

• Aged 18 years or older

RBC TRANSFUSION DOMAIN EXCLUSION CRITERIA:

* Contraindication to RBC transfusion (including known patient preference)
* Limitations of care put in place either through patient wishes or the treating medical teams.
* Participant has already received ECMO >12 hours. The start of ECMO is defined as the time of initiation of extracorporeal blood flow unless ECMO was initiated during a surgical intervention in which case the start of ECMO is defined as the arrival time into the initial ICU (post-surgery)
* The treating physician anticipates that ECMO treatment will cease before the end of tomorrow
* The treating physician deems the study is not in the patient's best interest
* The treating physician has concern regarding patient ability to tolerate restrictive or liberal transfusion trigger thresholds
* Actively listed for a solid organ transplant and has not yet received one
* Suspected or confirmed to be pregnant
* Previous ECMO treatment during the same hospital admission

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Daily Organ Support for patients on ECMO (DOSE-score). | 28-days.
  The primary outcome is the Daily Organ Support for patients on ECMO (DOSE-score), a 6-level daily ordinal outcome measured as the worst status of a patient on each day from day 1 through to day 28 inclusive, which reflects survival, organ support and resource utilisation:
  1. dead;
  2. on ECMO;
  3. invasively mechanically ventilated without ECMO;
  4. in ICU but not invasively mechanically ventilated nor on ECMO;
  5. in hospital; and
  6. discharged from the hospital alive.

SECONDARY OUTCOMES:
Development of major haemorrhage at 28 days | 28-days.
  Development of major haemorrhage
Development of intracranial haemorrhage at 28 days | 28 days
  Development of intracranial haemorrhage
Mortality at 28 days | 28 days
  Living status.
ECMO-free days at 28 days | 28 days
  Number of days not receiving ECMO
Ventilator-free days at 28 days | 28 days
  Number of days not receiving ventilation

OTHER OUTCOMES:
Mortality at 180 days | 180 days
  Platform Trial Tertiary Outcome
Disability at 180 days | 180 days
  Platform Trial Tertiary Outcome - measured by WHODAS 2.0 at 180-days
Functional Status at 180 days | 180 days
  Platform Trial Tertiary Outcome - measured using Lawton-Brody IADL and Barthel ADL
Quality of Life at 180 days | 180 days
  Platform Trial Tertiary Outcome - measured by Eq-5D-5L and EQ-VAS
ICU Length of Stay | 180 days
  Platform Trial Tertiary Outcome
Hospital Length of Stay | 180 days
  Platform Trial Tertiary Outcome - separated for survivors and non-survivors
Number and Nature of SAEs | 28 days
  RBC Transfusion Domain Specific Outcome
Mortality in ICU | 180 days
  RBC Transfusion Domain Specific Outcome
Total Blood Products | 28 days
  RBC Transfusion Domain Specific Outcome - administered until cessation of ECMO or 28 days, whichever occurs first
Total RBC Units | 28 days
  RBC Transfusion Domain Specific Outcome - administered until cessation of ECMO or 28 days, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, PhD FACP FAHMS, Study Chair — Monash University
Locations (3):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Hospital Sydney, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
No IPD is created as individual data are not shared. However, aggregated data presented in manuscripts and publications or similar works, will be accessible upon patient request or own investigation.